CLINICAL TRIAL: NCT01609283
Title: A Dose-escalation Safety Trial for Intrathecal Autologous Mesenchymal Stem Cell Therapy in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Anthony J. Windebank, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-008415
Record Dates: First submitted 2012-05-18; First posted 2012-05-31 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous Mesenchymal Stem Cells (Experimental)
  Interventions: Biological: autologous mesenchymal stem cells

INTERVENTIONS:
Biological: autologous mesenchymal stem cells — There will be five treatment groups of up to five patients each. Groups 1, 2 and 4 will receive a single dose of cells. Groups 3 and 5 will receive 2 doses of cells separated by one month. Intrathecal injections into new subjects will be timed so that there is a minimum of one week between subject injections. The cell dose per group is as follows:
  * Group 1: single intrathecal dose of 1 x 107 cells
  * Group 2: single intrathecal dose of 5 x 107 cells
  * Group 3: one intrathecal dose of 5 x 107 cells followed one month later by a second intrathecal dose of 5 x 107 cells
  * Group 4: single intrathecal dose of 1 x 108 cells
  * Group 5: one intrathecal dose of 1 x 108 cells followed one month later by a second intrathecal dose of 1 x 108 cells

SUMMARY:
The purpose of this study is to determine determine the safety of intraspinal delivery of mesenchymal stem cells (MSCs) to the cerebral spinal fluid of patients with Amyotrophic Lateral Sclerosis (ALS) using a dose-escalation study.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the safety of intrathecal delivery of autologous mesenchymal stem cells (MSCs) to the cerebrospinal fluid (CSF) of patients with ALS using a dose-escalation study. The trial will include 25 adult, non-ventilator-dependent patients with clinically definite amyotrophic lateral sclerosis (ALS). Cells will be isolated from adipose tissue, expanded ex vivo and then, after ~8 weeks, intrathecal (IT) autologous delivery of MSCs will be performed. There will be 5 treatment groups of up to 5 patients each. Groups 1, 2, and 4 will receive a single dose of cells. Groups 3 and 5 will receive 2 doses of cells separated by 1 month. Groups will be completed sequentially so that patients will not be enrolled into the next treatment group until at least 3 patients in the preceding group have completed the treatment and 1 month of additional observation without significant toxicity. All patients will be followed on a regular basis until death or for a minimum of 2 years after completion of the final infusion. Initial clinical follow-up will be weekly with scheduled blood, CSF and magnetic resonance imaging (MRI) evaluations. After 1 month, patients will have clinical evaluations at 3 month intervals, or earlier if indicated by clinical status.

Addendum: Five subjects from the Group 5 dosing level will received additional injections of MSCs in an extension of the original study, if tolerated.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have clinically-defined ALS as defined by the World Federation of Neurology criteria
* Age greater than 18 years
* If female, must be post-menopausal or had a hysterectomy
* Permanent resident or citizen of the United States
* History of a chronic onset of a progressive motor weakness of greater than one year, but less than two years duration
* Must have vital capacity greater than 65% of predicated for age, gender, and body type
* Able to comply with protocol requirements, including MRI testing
* Can provide written informed consent

Exclusion Criteria:

* Any clinically significant medical condition (e.g., within six months of baseline, had myocardial infarction, angina pectoris, and/or congestive heart failure) that, in the opinion of the investigator, would compromise the safety of patient.
* Autoimmunity, including Crohn's disease, rheumatoid arthritis, psoriasis
* Malignancy including melanoma with the exception of localized skin cancers (with no evidence of metastasis, significant invasion, or re-occurrence within three years of baseline). Any other malignancy will not be allowed.
* Active systemic or local infection near the lumbar puncture site
* Other active systemic disease as defined by laboratory abnormalities
* Use of herbal medications or other unapproved drugs
* Enrolled in an investigational drug trial within 30 days of baseline visit
* Kokmen Short Test of Mental Status score <32
* Beck's Depression Inventory score >18
* Presence of a tracheostomy
* Ventilator dependent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-05; Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicities | baseline -2 years after completion of the final infusion

SECONDARY OUTCOMES:
Number of patients with adverse events | baseline -2 years after completion of the final infusion
Change in serum sedimentation rate | baseline, 2 years after completion of the final infusion
Change in C-reactive protein levels | baseline, 2 years after completion of the final infusion
Change in complete blood counts | baseline, 2 years after completion of the final infusion
Change in total nucleated cell count in cerebrospinal fluid (CSF) | baseline, 2 years after completion of the final infusion
Change in protein level in cerebrospinal fluid (CSF) | baseline, 2 years after completion of the final infusion
Number of patients with presence of cancer cells in their cerebrospinal fluid (CSF) | baseline -2 years after completion of the final infusion

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Windebank, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camilleri ET, Gustafson MP, Dudakovic A, Riester SM, Garces CG, Paradise CR, Takai H, Karperien M, Cool S, Sampen HJ, Larson AN, Qu W, Smith J, Dietz AB, van Wijnen AJ. Identification and validation of multiple cell surface markers of clinical-grade adipose-derived mesenchymal stromal cells as novel release criteria for good manufacturing practice-compliant production. Stem Cell Res Ther. 2016 Aug 11;7(1):107. doi: 10.1186/s13287-016-0370-8. PMID 27515308
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials